CLINICAL TRIAL: NCT03176381
Title: Development of Tissue Predictors of Abiraterone Benefit in Men With mCRPC
Brief Title: Tissue Predictors of Abiraterone Benefit
Status: Completed | Type: Observational
Sponsor: Tianjin Medical University Second Hospital (Other)
Collaborators: Tianjin Medical University General Hospital (Other); Tianjin Medical University Cancer Institute and Hospital (Other); Beijing Chao Yang Hospital (Other); The Second Hospital of Hebei Medical University (Other); Affiliated Hospital of Hebei University (Other)
Responsible Party: Sponsor
Other Study IDs: mCRPC-PA
Record Dates: First submitted 2017-06-01; First posted 2017-06-05 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Metastatic Castration-resistant Prostate Cancer
Keywords: Prostatic Neoplasms; Abiraterone Acetate; FK506 binding protein 5; Neurotensin; yes-associated protein 1; AKR1C3 protein; Proliferating Cell Nuclear Antigen
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — RNA-seq with IHC of AKR1C3, FKB5 and PCNA were tested in the tissue specimen.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

SUMMARY:
This is an observational, prospective (study following participants forward in time), multi-center (study conducted in more than 1 center) study to identify the predictive factors that will effectively predict the response to abiraterone treatment in metastatic castration-resistant prostate cancer (mCRPC). The entire duration of study will be approximately 3 year. Participants will primarily be evaluated for achieving biochemical or radiological progression after receiving abiraterone treatment based on EAU 2017 practice guideline criteria. For this, we put our attentions on the HOXB3 (an alternative factor of WNT signaling pathway), FKBP5 (FK506 Binding Protein 5, Androgen-regulated gene), NTS (neurotensin, neuroendocrine differentiation can be induced by NTS) and YAP1 (yes-associated protein 1, a biomarker for cancer stem cell), which are selected from the data of gene-array for various subtypes of CRPC (unpublished data). Response to abiraterone treatment will also be predicted using other androgen-regulated genes like AKR1C3 and PCNA.

DETAILED DESCRIPTION:
It is now accepted that castration-resistant prostate cancer (CRPC) is not really androgen-independent and continues to rely on androgen signaling. Abiraterone is an inhibitor of cytochrome P450 17A1 (CYP17A1) that impairs androgen-receptor signaling by depleting adrenal and intratumoral androgens. After studies showed improved survival with abiraterone, it was approved by the Food and Drug Administration for the treatment of metastatic castration-resistant prostate cancer (mCRPC).

mCRPC is a syndrome other than a disease. The mechanisms of mCRPC contain aberrant activation of androgen signaling, abnormal transition between epithelial and mesenchymal and induction of neuroendocrine differentiation (NED). In addition, cellular heterogeneity represents an omnipresent feature in human tumors, which contain cells with diverse morphology, cytogenetic markers, growth kinetics, immunological characteristics, metastatic ability, and sensitivity to therapeutics.

This is an observational, prospective (study following participants forward in time), multi-center (study conducted in more than 1 center) study to identify the predictive factors that will effectively predict the response to abiraterone treatment in metastatic castration-resistant prostate cancer (mCRPC). The entire duration of study will be approximately 3 year. Participants will primarily be evaluated for achieving biochemical or radiological progression after receiving abiraterone treatment based on EAU 2017 practice guideline criteria. For this, we put our attentions on the FKBP5 (FK506 Binding Protein 5, Androgen-regulated gene), NTS (neurotensin, neuroendocrine differentiation can be induced by NTS) and YAP1 (yes-associated protein 1, a biomarker for cancer stem cell), which are selected from the data of gene-array for various subtypes of CRPC. Response to abiraterone treatment will also be predicted using other androgen-regulated genes like AKR1C3 and PCNA.

ELIGIBILITY:
Inclusion Criteria:

1. Participants who have given consent form;
2. Patients with a confirmed diagnosis of mCRPC according to EAU 2017 guideline;
3. Serum testosterone must reach castration level: <50 ng per deciliter;
4. Participants with life expectancy of at least 6 months based on the Investigator's clinical judgment.

Exclusion Criteria:

1. Participants who are allergic to contrast medium;
2. Patients were excluded if they planned to receive additional concurrent anticancer therapies;
3. Patients doesn't sign an informed consent form.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male only
Study Population: Participants having indication and planning to receiving abiraterone treatment.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2017-05-05 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
PSA response rates | 2 YEARS
  PSA response rates between FKBP5(protein)-positive and FKBP5(protein)-negative (including YAP1-positive and NTS-positive) patients; PSA response rates between patients with higher or lower expression of androgen-regulated genes (AKR1C3, FKB5, PCNA).

SECONDARY OUTCOMES:
PSA progression-free survival (pPFS) | 3 YEARS
  pPFS between FKBP5-positive and FKBP5-negative (including YAP1-positive and NTS-positive) patients; pPFS between patients with higher or lower expression of androgen-regulated genes (AKR1C3, FKB5, PCNA).
clinical or radiographic progression-free survival (cPFS) | 3 YEARS
  cPFS between FKBP5-positive and FKBP5-negative (including YAP1-positive and NTS-positive) patients; cPFS between patients with higher or lower expression of androgen-regulated genes (AKR1C3, FKB5, PCNA).
overall survival (OS) | 3 YEARS
  OS between FKBP5-positive and FKBP5-negative (including YAP1-positive and NTS-positive) patients; OS between patients with higher or lower expression of androgen-regulated genes (AKR1C3, FKB5, PCNA).

CONTACTS AND LOCATIONS:
Overall Officials: Rong Han, Principal Investigator — Tianjin Medical University Second Hospital
Locations (1):
- Tianjin Medical Unversity Second Hospital, Tianjin, China

IPD SHARING:
Plan to Share IPD: Yes
IPD can be got by contacting researchers

REFERENCES:
- [Background] Longo DL. New therapies for castration-resistant prostate cancer. N Engl J Med. 2010 Jul 29;363(5):479-81. doi: 10.1056/NEJMe1006300. No abstract available. PMID 20818868
- [Background] Ryan CJ, Tindall DJ. Androgen receptor rediscovered: the new biology and targeting the androgen receptor therapeutically. J Clin Oncol. 2011 Sep 20;29(27):3651-8. doi: 10.1200/JCO.2011.35.2005. Epub 2011 Aug 22. PMID 21859989
- [Background] O'Donnell A, Judson I, Dowsett M, Raynaud F, Dearnaley D, Mason M, Harland S, Robbins A, Halbert G, Nutley B, Jarman M. Hormonal impact of the 17alpha-hydroxylase/C(17,20)-lyase inhibitor abiraterone acetate (CB7630) in patients with prostate cancer. Br J Cancer. 2004 Jun 14;90(12):2317-25. doi: 10.1038/sj.bjc.6601879. PMID 15150570
- [Background] Attard G, Reid AH, Yap TA, Raynaud F, Dowsett M, Settatree S, Barrett M, Parker C, Martins V, Folkerd E, Clark J, Cooper CS, Kaye SB, Dearnaley D, Lee G, de Bono JS. Phase I clinical trial of a selective inhibitor of CYP17, abiraterone acetate, confirms that castration-resistant prostate cancer commonly remains hormone driven. J Clin Oncol. 2008 Oct 1;26(28):4563-71. doi: 10.1200/JCO.2007.15.9749. Epub 2008 Jul 21. PMID 18645193
- [Background] Scher HI, Fizazi K, Saad F, Taplin ME, Sternberg CN, Miller K, de Wit R, Mulders P, Chi KN, Shore ND, Armstrong AJ, Flaig TW, Flechon A, Mainwaring P, Fleming M, Hainsworth JD, Hirmand M, Selby B, Seely L, de Bono JS; AFFIRM Investigators. Increased survival with enzalutamide in prostate cancer after chemotherapy. N Engl J Med. 2012 Sep 27;367(13):1187-97. doi: 10.1056/NEJMoa1207506. Epub 2012 Aug 15. PMID 22894553
- [Background] de Bono JS, Logothetis CJ, Molina A, Fizazi K, North S, Chu L, Chi KN, Jones RJ, Goodman OB Jr, Saad F, Staffurth JN, Mainwaring P, Harland S, Flaig TW, Hutson TE, Cheng T, Patterson H, Hainsworth JD, Ryan CJ, Sternberg CN, Ellard SL, Flechon A, Saleh M, Scholz M, Efstathiou E, Zivi A, Bianchini D, Loriot Y, Chieffo N, Kheoh T, Haqq CM, Scher HI; COU-AA-301 Investigators. Abiraterone and increased survival in metastatic prostate cancer. N Engl J Med. 2011 May 26;364(21):1995-2005. doi: 10.1056/NEJMoa1014618. PMID 21612468
- [Background] Ryan CJ, Smith MR, de Bono JS, Molina A, Logothetis CJ, de Souza P, Fizazi K, Mainwaring P, Piulats JM, Ng S, Carles J, Mulders PF, Basch E, Small EJ, Saad F, Schrijvers D, Van Poppel H, Mukherjee SD, Suttmann H, Gerritsen WR, Flaig TW, George DJ, Yu EY, Efstathiou E, Pantuck A, Winquist E, Higano CS, Taplin ME, Park Y, Kheoh T, Griffin T, Scher HI, Rathkopf DE; COU-AA-302 Investigators. Abiraterone in metastatic prostate cancer without previous chemotherapy. N Engl J Med. 2013 Jan 10;368(2):138-48. doi: 10.1056/NEJMoa1209096. Epub 2012 Dec 10. PMID 23228172
- [Background] Tang DG. Understanding cancer stem cell heterogeneity and plasticity. Cell Res. 2012 Mar;22(3):457-72. doi: 10.1038/cr.2012.13. Epub 2012 Jan 17. PMID 22357481
- [Background] Mulholland DJ, Tran LM, Li Y, Cai H, Morim A, Wang S, Plaisier S, Garraway IP, Huang J, Graeber TG, Wu H. Cell autonomous role of PTEN in regulating castration-resistant prostate cancer growth. Cancer Cell. 2011 Jun 14;19(6):792-804. doi: 10.1016/j.ccr.2011.05.006. Epub 2011 May 27. PMID 21620777
- [Background] Swift SL, Burns JE, Maitland NJ. Altered expression of neurotensin receptors is associated with the differentiation state of prostate cancer. Cancer Res. 2010 Jan 1;70(1):347-56. doi: 10.1158/0008-5472.CAN-09-1252. PMID 20048080
- [Background] Valerie NC, Casarez EV, Dasilva JO, Dunlap-Brown ME, Parsons SJ, Amorino GP, Dziegielewski J. Inhibition of neurotensin receptor 1 selectively sensitizes prostate cancer to ionizing radiation. Cancer Res. 2011 Nov 1;71(21):6817-26. doi: 10.1158/0008-5472.CAN-11-1646. Epub 2011 Sep 8. PMID 21903767
- [Background] Selth LA, Das R, Townley SL, Coutinho I, Hanson AR, Centenera MM, Stylianou N, Sweeney K, Soekmadji C, Jovanovic L, Nelson CC, Zoubeidi A, Butler LM, Goodall GJ, Hollier BG, Gregory PA, Tilley WD. A ZEB1-miR-375-YAP1 pathway regulates epithelial plasticity in prostate cancer. Oncogene. 2017 Jan 5;36(1):24-34. doi: 10.1038/onc.2016.185. Epub 2016 Jun 6. PMID 27270433
- [Background] Thoma C. Prostate cancer: Targetable YAP1-AR interaction key to disease progression. Nat Rev Urol. 2015 Nov;12(11):596. doi: 10.1038/nrurol.2015.240. Epub 2015 Sep 22. No abstract available. PMID 26390969